CLINICAL TRIAL: NCT02259634
Title: Impact of Patient Navigators on Health Education and Quality of Life in Formerly Incarcerated Patients
Brief Title: Study on the Impact of Patient Navigators on the Health Education and Quality of Life in Formerly Incarcerated Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Target sample size not reached for enrollment.
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Hunter College of The City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AD-1304-6854
Record Dates: First submitted 2014-09-15; First posted 2014-10-08 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: HIV/AIDS; Diabetes Mellitus; Hypertension; Substance Use
Keywords: Patient Navigation; Motivational Interviewing; Formerly Incarcerated; Health Education; Quality of Life; Healthcare Utilization
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diabetes Mellitus; Hypertension; Substance-Related Disorders; Health Education | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Navigation (Experimental): Intensive Patient Navigation with Motivational Interviewing and Health Education for 8 months 18 month follow-up
  Interventions: Behavioral: Patient Navigation
- Treatment as Usual (No Intervention): Case Management and Medical Care as provided by the Coming Home Program at Mount Sinai St. Luke's Institute of Advanced Medicine, Morningside Clinic

INTERVENTIONS:
Behavioral: Patient Navigation — Motivational Interviewing
  Arms: Patient Navigation

SUMMARY:
This is a 3-year prospective randomized comparative study of the efficacy of patient navigation on health education, health related quality of life, healthcare utilization, and medical outcomes in formerly incarcerated individuals. Individuals will be randomized to the patient-navigator intervention or to a care-as-usual control condition. A total of 300 recently incarcerated individuals will be enrolled with 150 subjects each in the intervention and usual care group.

The investigators hypothesize that the intervention will improve health education, health related quality of life, adherence to clinical appointments, glycemic/blood pressure control, and virologic suppression in HIV-infected. The results of this study will demonstrate interventions to eliminate health disparities in a highly marginalized group going through the transitional phase of re-entry into the community.

DETAILED DESCRIPTION:
This is a 3-year prospective randomized comparative trial that will examine the impact of an intervention that incorporates peer navigators to improve health education (heiQ), health related quality of life (HRQOL-14), healthcare utilization, and medical outcomes compared to usual care among formerly incarcerated individuals as they transition from the correctional system into the community over the course of 18 months. Multiple studies have shown the efficacy of patient navigators in improving healthcare utilization and outcomes in marginalized populations, but neither intervention has been studied with the formerly incarcerated population. A total of 300 formerly incarcerated individuals will be enrolled into the trial. This intervention is inherently patient-centered, as it facilitates a process by which patients continuously define and shape their engagement with the health care system. The potential impact of the study findings include: 1) evidence for or against the use of patient navigators to enhance linkage and engagement into care; 2) health outcomes that either support or discourage the use of patient navigators with formerly incarcerated people; 3) expansion of knowledge to inform the development of targeted interventions for this vulnerable population; and 4) dissemination of results that may contribute to larger scale studies that can be implemented widely with the aim at eliminating health disparities in a highly marginalized group of people. The investigators specific aim is to conduct a randomized comparative trial that will provide the evidence base to address two primary research questions:

1. How does the use of patient navigators impact health education and health related quality of life of individuals as they transition from the correctional system into the community?
2. How does a patient navigator for formerly incarcerated patients improve metrics of health care utilization (adherence to medical appointments, fewer visits to emergency rooms) and health outcomes (glycemic index, blood pressure control, and/or virological suppression in HIV-infected) compared to usual care of automated appointment reminder phone calls?

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* English or Spanish speaking
* release from the correctional system within the previous 6 months

Exclusion Criteria:

* unable to provide informed consent
* report duration of incarceration of less than 5 days
* report history of incarceration more than 6 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Health Education Impact | 18 months
  Health education impact questionnaire (heiQ)
Quality of Life | 18 months
  Health related quality of life (HRQOL-14)

SECONDARY OUTCOMES:
Health Outcomes | 18 months
  Glycemic index, blood pressure control, and/or virological suppression in HIV-infected
Healthcare Utilization | 18 months
  Adherence to clinical appointments and contact with emergency services (emergency department)

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Osorio, MD, MPH, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (2):
- United States (2):
  - Mount Sinai St. Luke's, New York, New York
  - Hunter College at The City University of New York, New York, New York